CLINICAL TRIAL: NCT01470014
Title: Cardiac Computed Tomography: Characteristics of Isolated Left Ventricular Non-compaction
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK 2011-0099
Record Dates: First submitted 2011-10-27; First posted 2011-11-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Left Ventricular Noncompaction; Isolated Noncompaction of the Ventricular Myocardium
Keywords: isolated left ventricular non-compaction; cardiac computed tomography; cardiac magnet resonance imaging; echocardiography
MeSH Terms: conditions — Isolated Noncompaction of the Ventricular Myocardium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- IVNC
- differential diagnosis to IVNC

SUMMARY:
The diagnostic criteria for isolated left ventricular non-compaction cardiomyopathy (IVNC) have been well established for echocardiography and cardiac magnetic resonance, such validation is lacking for computed tomography (CT). Such criteria are of great clinical relevance as a growing number of patients undergo a cardiac CT scan in daily clinical routine.

The investigators aim to test the diagnostic accuracy of cardiac CT in distinguishing IVNC from lesser degrees of trabecular layering seen in potential differential diagnoses such as cardiomyopathies and left ventricular hypertrophy or dilation.

The investigators hypothesize that echocardiographic diagnosed pathological trabeculation can be distinguished by determining the ratio of non-compacted to compacted myocardium on cardiac CT.

ELIGIBILITY:
Inclusion criteria:

* Established diagnosis of IVNC or differential diagnosis
* Age: Men > 30 years, women > 50 years without menstruation for at least 2 month.
* Written informed consent to participate

Exclusion criteria: Contraindication for cardiac CT

* Renal insufficiency (GFR < 60ml/min)
* Known allergy to iodinated contrast agent
* Known Hyperthyroidism
* Non-sinus rhythm
* Known premature ventricular or supraventricular beats
* Hypotension (systolic blood pressure < 100mmHg)

Contraindication for CMR

* Implanted cardiac pacemaker or defibrillator
* Other implanted medical devices (e.g. implantable cardioverter-defibrillator)
* Claustrophobia
* Known premature ventricular or supraventricular beats
* Pregnancy
* Claustrophobia

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Department of Cardiology and Cardiac Imaging Division. They will be asked if they want to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Tanner, Prof. MD, Principal Investigator — University Hospital Zurich, Division of Cardiology
Locations (1):
- Zurich, Switzerland